CLINICAL TRIAL: NCT03490539
Title: Prospective Multicenter Observational Cohort Study of Comparative Effectiveness of Disease-modifying Treatments for Myasthenia Gravis
Brief Title: Disease-Modifying Treatments for Myasthenia Gravis
Acronym: PROMISE-MG
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00087883
Record Dates: First submitted 2018-03-21; First posted 2018-04-06 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Neurological Disorder; Autoimmune Diseases
Keywords: observational; comparative effectiveness; myasthenia gravis
MeSH Terms: conditions — Nervous System Diseases; Autoimmune Diseases; Myasthenia Gravis | interventions — Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- azathioprine (AZT): Patients with MG who are receiving azathioprine as part of routine clinical care
  Interventions: Drug: Azathioprine
- mycophenolate mofetil (MMF): Patients with MG who are receiving mycophenolate mofetil as part of routine clinical care
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — oral tablets
  Other Names: Cellcept
  Groups: mycophenolate mofetil (MMF)
Drug: Azathioprine — oral tablet
  Other Names: Imuran
  Groups: azathioprine (AZT)

SUMMARY:
This study is designed to address the evidence gaps in a real-world setting and help patients with MG choose treatments that are best suited to them. It is a prospective, multicenter observational cohort study of comparative effectiveness of MG treatments, with a patient-centered primary outcome measure, to guide clinicians, patients and payers regarding the choice of treatment options for this chronic and serious disease.

Primary: To compare the effectiveness of azathioprine (AZT) and mycophenolate mofetil (MMF).

Secondary: To compare the outcomes in patients receiving an adequate dose and duration of AZT or MMF over the 2-3 year study period, vs. patients not receiving adequate doses and duration of these agents

DETAILED DESCRIPTION:
Design & procedures - This is an observational study in the real world clinical setting to evaluate immunosuppressive treatment (IS) of myasthenia gravis (MG). Patients with acquired autoimmune MG ≥ 18 years of age who are not on IS agents, and have not been on corticosteroids for at least 30 days will be enrolled at 20 sites in the US and Canada. These patients will be treated according to the physician's judgment and patient preferences as in routine clinical practice. Patients will be followed prospectively, with the frequency of clinical visits and laboratory monitoring determined by the treating physician, which may differ among patients. Standard outcome measures measuring efficacy and adverse effects that are used in clinical practice will be collected, with emphasis on patient reported outcomes. Informed consent will be obtained using an approved consent form. Patient identifiable / clinical information from the medical record, including the study outcome measures will be uploaded to a centralized REDCap database. The investigators plan to recruit 220 patients, adjusting for a 10% drop out rate, with a final sample of 200 patients for analysis.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study must fulfill all of the following criteria:

1. Age ≥ 18 years of age
2. Acquired autoimmune MG, with weakness and confirmed by one or more of the following:

   1. Elevated AChR or MuSK antibodies
   2. Unequivocal response to cholinesterase inhibitors
   3. Abnormal RNS or increased jitter (without nerve or muscle disease sufficient to produce a decrement or increased jitter)
3. Patients seen initially at the participating center after January 1, 2017.
4. Patients on pyridostigmine at the first evaluation at the participating center ("baseline visit") may be included if pyridostigmine was started ≤3 months before the baseline visit.
5. Patients who received corticosteroids >90 days prior to baseline visit for a non-MG indication may be included. (Patients who have received corticosteroids for a non-MG indication between 31 and 90 days before baseline visit will be evaluated by the primary investigators on a case by case basis to determine if the extent and dose of corticosteroid could have impacted the course of MG or symptoms of MG.)

Exclusion Criteria:

Patients fulfilling any of the following criteria are not eligible for inclusion in this study. No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible participants.

1. Patients with non-autoimmune MG (congenital myasthenic syndromes, drug-induced MG)
2. Patients on immunosuppressive agents at the baseline visit.
3. Patients who have previously received steroids for the treatment of MG.
4. Patients with steroid use for a non-MG indication < 30 days prior to the baseline visit.
5. Patients with previous thymectomy, IVIg or plasma exchange, or treatment with a non-steroidal immunosuppressive agent (azathioprine, mycophenolate mofetil cyclosporine, methotrexate, cyclophosphamide, tacrolimus, rituximab, or any investigational immunosuppressive agent). Patients who have outcomes measured within 24 hours after initiation of IVIg or PLEX are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MG patients with autoimmune MG
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Change in Patient-Reported Myasthenia Gravis Quality of Life, 15, revised ( MG-QOL15r) | Baseline, 24-36 months
  Measures MG symptoms, physical, social and emotional functioning related to MG, with 15 items, 3 response option, 0-2 for each item, Total score range 0-30, higher scores indicating worse function
Change in composite outcome of clinical improvement and adverse effects | Baseline, 24-36 months
  measured by a composite of clinical improvement and adverse effects of treatments. Clinical improvement: achievement of MGFA Post-Intervention Status (PIS) Minimal Manifestation Status (MM) or better, defined below.
  Adverse effects end point: no more than Grade 1 CTCAE (Common Terminology Criteria for Adverse Events) medication side-effects, defined below.
  MGFA PIS- MM: the patient has no symptoms or functional limitations from MG but has some weakness on examination of some muscles
  CTCAE: list of adverse event (AE) terms commonly encountered in oncology but is useful to monitor the side effects of any intervention Each AE term is defined and graded on a 1 to 5 scale indicating the severity of the AE, 1 representing the mildest side effect and 5 representing death Grade 1 CTCAE side-effects: "asymptomatic or only mild symptoms; intervention not indicated"

SECONDARY OUTCOMES:
Change in Myasthenia gravis composite (MGC) scores | Baseline, 24-36 months
  10 item scale of patient-reported functions and clinician-reported examination findings.
  Scores range from 0-50 (0- normal and 50- most severe)
Change in Myasthenia Gravis Activities of Daily Living Scale (MG-ADL) | Baseline, 24-36 months
  Patient-reported 8- item questionnaire evaluating commonly reported symptoms in MG on a 4 response scale from 0-3 (0 - normal, 3- highest disability) Range 0-24, higher score is worse
Change in Myasthenia Gravis Manual Muscle Test scores (MG-MMT) | Baseline, 24-36 months
  Clinician-assessed scale of 18 muscle functions commonly affected by MG, each graded from 0 (normal) to 4 (paralyzed/unable to perform), Range 0-120, higher score reflects worse function
Change in Visual Analogue Scale (VAS) for Disease Severity | Baseline, 24-36 months
  Patient perception of disease severity measured in millimeters on a 100 mm line. Higher number indicates more severe disease
Change in Visual Analogue Scale (VAS) for Treatment Side effects | Baseline, 24-36 months
  patient perception of side effects of treatment measured in millimeters on a 100 mm line. Higher number indicates worse side effects
Change in number of hospitalizations for MG | Baseline, 24-36 months
  counts of hospitalizations for MG- higher count is worse

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Guptill, MD, Principal Investigator — Duke University; Donald Sanders, MD, Principal Investigator — Duke University; Pushpa Narayanaswami, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (19):
- United States (17):
  - Stanford University, Palo Alto, California
  - Unversity of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - University at Buffalo, SUNY, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Vermont - Larner College of Medicine, Burlington, Vermont
- Canada (2):
  - University of Alberta Hospital, Faculty of Medicine, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deenen JC, Horlings CG, Verschuuren JJ, Verbeek AL, van Engelen BG. The Epidemiology of Neuromuscular Disorders: A Comprehensive Overview of the Literature. J Neuromuscul Dis. 2015;2(1):73-85. PMID 28198707
- [Background] Sanders DB, Wolfe GI, Narayanaswami P. Author response: International consensus guidance for management of myasthenia gravis: Executive summary. Neurology. 2017 Jan 31;88(5):505-506. doi: 10.1212/WNL.0000000000003570. No abstract available. PMID 28138082
- [Background] Burns TM, Sadjadi R, Utsugisawa K, Gwathmey KG, Joshi A, Jones S, Bril V, Barnett C, Guptill JT, Sanders DB, Hobson-Webb L, Juel VC, Massey J, Gable KL, Silvestri NJ, Wolfe G, Cutter G, Nagane Y, Murai H, Masuda M, Farrugia ME, Carmichael C, Birnbaum S, Hogrel JY, Nafissi S, Fatehi F, Ou C, Liu W, Conaway M. International clinimetric evaluation of the MG-QOL15, resulting in slight revision and subsequent validation of the MG-QOL15r. Muscle Nerve. 2016 Dec;54(6):1015-1022. doi: 10.1002/mus.25198. Epub 2016 Nov 7. PMID 27220659
- [Background] Mullins LL, Carpentier MY, Paul RH, Sanders DB; Muscle Study Group. Disease-specific measure of quality of life for myasthenia gravis. Muscle Nerve. 2008 Aug;38(2):947-56. doi: 10.1002/mus.21016. PMID 18697209
- [Background] Burns TM, Grouse CK, Wolfe GI, Conaway MR, Sanders DB; MG Composite and MG-OL15 Study Group. The MG-QOL15 for following the health-related quality of life of patients with myasthenia gravis. Muscle Nerve. 2011 Jan;43(1):14-8. doi: 10.1002/mus.21883. PMID 21082698
- [Background] Jaretzki A 3rd, Barohn RJ, Ernstoff RM, Kaminski HJ, Keesey JC, Penn AS, Sanders DB. Myasthenia gravis: recommendations for clinical research standards. Task Force of the Medical Scientific Advisory Board of the Myasthenia Gravis Foundation of America. Neurology. 2000 Jul 12;55(1):16-23. doi: 10.1212/wnl.55.1.16. No abstract available. PMID 10891897
- [Background] Burns TM, Conaway M, Sanders DB; MG Composite and MG-QOL15 Study Group. The MG Composite: A valid and reliable outcome measure for myasthenia gravis. Neurology. 2010 May 4;74(18):1434-40. doi: 10.1212/WNL.0b013e3181dc1b1e. PMID 20439845
- [Background] Sadjadi R, Conaway M, Cutter G, Sanders DB, Burns TM; MG Composite MG-QOL15 Study Group. Psychometric evaluation of the myasthenia gravis composite using Rasch analysis. Muscle Nerve. 2012 Jun;45(6):820-5. doi: 10.1002/mus.23260. PMID 22581534
- [Background] Burns TM, Conaway MR, Cutter GR, Sanders DB; Muscle Study Group. Construction of an efficient evaluative instrument for myasthenia gravis: the MG composite. Muscle Nerve. 2008 Dec;38(6):1553-62. doi: 10.1002/mus.21185. PMID 19016543
- [Background] Wolfe GI, Herbelin L, Nations SP, Foster B, Bryan WW, Barohn RJ. Myasthenia gravis activities of daily living profile. Neurology. 1999 Apr 22;52(7):1487-9. doi: 10.1212/wnl.52.7.1487. PMID 10227640
- [Background] Sanders DB, Tucker-Lipscomb B, Massey JM. A simple manual muscle test for myasthenia gravis: validation and comparison with the QMG score. Ann N Y Acad Sci. 2003 Sep;998:440-4. doi: 10.1196/annals.1254.057. No abstract available. PMID 14592912
- [Background] Gilhus NE, Verschuuren JJ. Myasthenia gravis: subgroup classification and therapeutic strategies. Lancet Neurol. 2015 Oct;14(10):1023-36. doi: 10.1016/S1474-4422(15)00145-3. PMID 26376969
- [Background] Bang H, Robins JM. Doubly robust estimation in missing data and causal inference models. Biometrics. 2005 Dec;61(4):962-73. doi: 10.1111/j.1541-0420.2005.00377.x. PMID 16401269
- [Background] Li F, Morgan KL, Zaslavsky AM. Balancing Covariates via Propensity Score Weighting. Journal of the American Statistical Association 2016;(In press).
- [Background] Crump RK. Dealing with limited overlap in estimation of average treatment effects. Biometrika 2009;96(1):187-199.
- [Background] Meriggioli MN, Sanders DB. Disorders of Neuromuscular Transmission. In: Bradley WG, Daroff RB, Fenichel GM, Jankovic J, Mazziotta JC, editors. Neurology in Clinical Practice. 6 ed. Philadelphia: Elsevier/Saunders; 2012. p 2046-2065.
- [Derived] Narayanaswami P, Sanders DB, Thomas L, Thibault D, Blevins J, Desai R, Krueger A, Bibeau K, Liu B, Guptill JT; PROMISE-MG Study Group. Comparative effectiveness of azathioprine and mycophenolate mofetil for myasthenia gravis (PROMISE-MG): a prospective cohort study. Lancet Neurol. 2024 Mar;23(3):267-276. doi: 10.1016/S1474-4422(24)00028-0. PMID 38365379
- See also: U.S. Department of Health and Human Services. Common Terminology Criteria for Adverse Events (CTCAE) v 4.03 — https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/